CLINICAL TRIAL: NCT00968721
Title: Decisional Influences and IBD Patients' Medication Use
Brief Title: Decisional Influences and Inflammatory Bowel Disease (IBD) Patients' Medication Use
Status: Terminated | Type: Observational
Why Stopped: lack of support
Sponsor: Vanderbilt University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 090527
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Inflammatory bowel disease; Crohn's disease; Ulcerative colitis; medication adherence; Decisional influences
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD patients

SUMMARY:
The primary purpose of this study is to pilot test an instrument that the investigators will develop to assess decision influences on inflammatory bowel disease patients' medication adherence decision-making.

This pilot study will use an exploratory, descriptive cross-sectional survey approach to pilot test the instrument and answer the research questions.

The main hypothesis is that patients at risk for intentionally modifying their prescribed medication regimen will differ on influences on decision-making, health status, and utilization of the IBD clinic services compared to those who are intentionally adherent and who continue adherence over time.

DETAILED DESCRIPTION:
Clinical research has produced significant advances in the pharmacologic management of inflammatory bowel disease (IBD). Preliminary research, however, suggest that patient non-adherence may be blunting medication effectiveness. The etiology of medication non-adherence likely depends on several coexisting factors. We believe that naturalistic decision making links patient level/ "micro" variables to services-level/ "macro" variables and behavioral outcomes. Every day, natural decisions about medication use are likely made in the context of patients' experience of their illness, knowledge about the illness and treatments, the physician-patient relationship, personal priorities and values, and other influences related to deciding to use medicine. By their very nature, illness related decisions are uncertain and risky because outcomes are unknown and patients often have limited knowledge and experience of the progression of their chronic illness. During the progression of an illness, patients may experiment with and analyze risks and benefits of therapies and relying on interpersonal interaction with health-care professionals to determine the self-management strategies best suited to patients and their life goals. Patient decision-making is thus and iterative process that evolves over time. An understanding of medication use decisions requires the description and understanding of those decision influences that may affect medication use decision-making over the course of the illness. Therefore, the primary purpose of this study is to develop and test a psychometric instrument that assesses influences on patients' decisions to use/not use their IBD medication.

The main hypothesis underlying the instrument development project is that patients at risk for intentionally modifying their prescribed medication regimen will differ on influences on decision-making, health status, and utilization of the IBD clinic services compared to those who are intentionally adherent and who continue adherence over time.

The following questions will be studied:

* What influences do therapeutic values, task difficulty, physician-patient relationship, information sources, personal beliefs and values have on patients' IBd medication adherence?
* What are the relationships between decision influences and illness activity?
* What associations exist among decision influences, illness activity, medication adherence and utilization of IBD Clinic services?

ELIGIBILITY:
Inclusion Criteria:

* All Vanderbilt University Medical Center IBD patients that are 18 years or older
* Those who volunteered to participate in this online web-based survey study.

Exclusion Criteria:

* Vanderbilt University Medical Center patients unable to take the survey because they do not have an e-mail address or access to one.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Vanderbilt University Medical Center Research Recruitment Registry will be used to identify the medical record and phone numbers of all VUMC patients recieving treatment for IBD.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
What influences do therapeutic values, task difficulty, physician-patient relationship, information sources, personal beliefs and values have on patients' IBd medication adherence? | 1 year

SECONDARY OUTCOMES:
What are the relationships between decision influences and illness activity? | 1 year
What associations exist among decision influences, illness activity, medication adherence and utilization of IBD Clinic services? | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Gaines, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Inflammatory Bowel Disease Clinic c/o Divison of Gastroenterology, Hepatology and Nutrition, Department of Medicine, School of Medicine, Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Cerveny P, Bortlik M, Kubena A, Vlcek J, Lakatos PL, Lukas M. Nonadherence in inflammatory bowel disease: results of factor analysis. Inflamm Bowel Dis. 2007 Oct;13(10):1244-9. doi: 10.1002/ibd.20189. PMID 17538983
- [Background] Ediger JP, Walker JR, Graff L, Lix L, Clara I, Rawsthorne P, Rogala L, Miller N, McPhail C, Deering K, Bernstein CN. Predictors of medication adherence in inflammatory bowel disease. Am J Gastroenterol. 2007 Jul;102(7):1417-26. doi: 10.1111/j.1572-0241.2007.01212.x. Epub 2007 Apr 16. PMID 17437505
- [Background] Harvey RF, Bradshaw JM. A simple index of Crohn's-disease activity. Lancet. 1980 Mar 8;1(8167):514. doi: 10.1016/s0140-6736(80)92767-1. No abstract available. PMID 6102236
- [Background] Hicks FD, Holm K. Self-management decision influences in heart failure: a preliminary investigation. Clin Nurs Res. 2003 Feb;12(1):69-84. doi: 10.1177/1054773803238741. PMID 12583500
- [Background] Horne, R. The medication adherence report scale. University of Brighton, Brighton, UK, 2004.
- [Background] Johnson MJ. The Medication Adherence Model: a guide for assessing medication taking. Res Theory Nurs Pract. 2002 Fall;16(3):179-92. doi: 10.1891/rtnp.16.3.179.53008. PMID 12472293
- [Background] Kane SV, Brixner D, Rubin DT, Sewitch MJ. The challenge of compliance and persistence: focus on ulcerative colitis. J Manag Care Pharm. 2008 Jan;14(1 Suppl A):s2-12; quiz s13-5. doi: 10.18553/jmcp.2008.14.s1-a.1a. PMID 18240888
- [Background] Kane SV, Loftus EV Jr, Dubinsky MC, Sederman R. Disease perceptions among people with Crohn's disease. Inflamm Bowel Dis. 2008 Aug;14(8):1097-101. doi: 10.1002/ibd.20418. PMID 18338774
- [Background] Riegel B, Carlson B, Moser DK, Sebern M, Hicks FD, Roland V. Psychometric testing of the self-care of heart failure index. J Card Fail. 2004 Aug;10(4):350-60. doi: 10.1016/j.cardfail.2003.12.001. PMID 15309704
- [Background] Sewitch MJ, Abrahamowicz M, Dobkin PL, Tamblyn R. Measuring differences between patients' and physicians' health perceptions: the patient-physician discordance scale. J Behav Med. 2003 Jun;26(3):245-64. doi: 10.1023/a:1023412604715. PMID 12845937
- [Background] Sewitch MJ, Abrahamowicz M, Barkun A, Bitton A, Wild GE, Cohen A, Dobkin PL. Patient nonadherence to medication in inflammatory bowel disease. Am J Gastroenterol. 2003 Jul;98(7):1535-44. doi: 10.1111/j.1572-0241.2003.07522.x. PMID 12873575
- [Background] Powell-Tuck J, Bown RL, Lennard-Jones JE. A comparison of oral prednisolone given as single or multiple daily doses for active proctocolitis. Scand J Gastroenterol. 1978;13(7):833-7. doi: 10.3109/00365527809182199. PMID 364626
- [Background] Wroe AL. Intentional and unintentional nonadherence: a study of decision making. J Behav Med. 2002 Aug;25(4):355-72. doi: 10.1023/a:1015866415552. PMID 12136497